CLINICAL TRIAL: NCT00348881
Title: Large Scale Safety and Immunogenicity Study of a DTaP-Hep B-PRP-T Combined Vaccine Compared to Tritanrix HepB/Hib™, Both Given Concomitantly With OPV at 6, 10, and 14 Weeks of Age in Healthy Filipino Infants
Brief Title: Study Comparing a DTaP-HB-PRP~T Combined Vaccine With Tritanrix HepB/Hib™, Concomitantly With OPV in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AL201
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-08

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Influenza
Keywords: Diphtheria; Tetanus; Pertussis; Hepatitis B Hansenula (HB); Haemophilus influenzae type b
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Influenza, Human; Haemophilus Infections | interventions — Poliovirus Vaccine, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: DTaP-Hep B-PRP-T + OPV vaccine (Experimental): Participants received 3 doses of the DTaP-Hep B-PRP-T concomitantly with OPV vaccine, 1 dose each at 6, 10, and 14 weeks of age.
  Interventions: Biological: DTaP-HB-PRP~T combined vaccine; Biological: Oral poliomyelitis vaccine (OPV)
- Group 2: Tritanrix-HepB/Hib™ + OPV vaccine (Active Comparator): Participants received 3 doses of the Tritanrix-HepB/Hib™ concomitantly with OPV vaccine, 1 dose each at 6, 10, and 14 weeks of age.
  Interventions: Biological: Tritanrix-HepB/Hib™ vaccine; Biological: Oral poliomyelitis vaccine (OPV)

INTERVENTIONS:
Biological: DTaP-HB-PRP~T combined vaccine — 0.5 mL, Intramuscular
  Arms: Group 1: DTaP-Hep B-PRP-T + OPV vaccine
Biological: Tritanrix-HepB/Hib™ vaccine — 0.5 mL, Intramuscular
  Arms: Group 2: Tritanrix-HepB/Hib™ + OPV vaccine
Biological: Oral poliomyelitis vaccine (OPV) — Oral co-administered with study vaccine.

SUMMARY:
This is a study to compare the safety and immune response of a pentavalent DTaP-HB-PRP~T combined vaccine with Tritanrix-HepB/Hib™, when both are given concomitantly with OPV at 6, 10, and 14 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

At Screening:

* 0 to 3 day old infants
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg
* Apgar score ≥ 7 at three minutes after birth
* Informed consent form signed by one parent or legal representative if appropriate (independent witness mandatory if parent is illiterate)

At Inclusion:

* Six weeks of age
* Received a dose of Hepatitis B (HB) in the first three days of life
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

At Screening:

* Illness at a stage that could interfere with trial conduct or completion
* Any vaccination before HB vaccination (except bacille Calmette-Guérin [BCG] given at birth)
* Vaccination planned in the 4 to 6 weeks following the first trial vaccination (except BCG if not given at birth)
* Acute illness on the day of screening.

At Screening and at Inclusion:

* Blood or blood-derived products received since birth
* Planned participation in another clinical trial during the present trial period
* Mother known as seropositive to Human immunodeficiency virus (HIV) or Hepatitis C, or as carrying the HB surface antigen (HBsAg)
* Known thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination
* Known hypersensitivity to any component of any vaccine to be used in the trial (including neomycin and polymixin B)

At Inclusion:

* Non-trial vaccine administered since birth, except Bacille Calmette-Guérin (BCG)
* Participation in another clinical trial before the first trial vaccination
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroid therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Vaccination other than with the study vaccines planned in the 12 weeks following inclusion
* Documented history of pertussis, tetanus, diphtheria, polio, H. influenza type b, or HB infection (confirmed clinically, serologically, or microbiologically)
* History of seizures
* Febrile (rectal temperature ≥ 38.0°C) or acute illness on the day of inclusion.

Ages: 42 Days to 50 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2133 (Actual)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- Philippines (4):
  - Alabang, Muntinlupa City
  - Putatan, Muntinlupa City
  - Tunasan, Muntinlupa City
  - Filinvest, Corporate City

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 17 May 2006 to 26 September 2006 in 1 clinic center in the Philippines.
Pre-assignment Details: A total of 2133 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received 3 doses of the DTaP-Hep B-PRP-T concomitantly with oral poliomyelitis vaccine (OPV), 1 dose each at 6, 10, and 14 weeks of age.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received 3 doses of Tritanrix-Hep B/ Hib™ concomitantly with oral poliomyelitis vaccine (OPV) at 6, 10 and 14 weeks of age.
Period: Overall Study
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Started | 1424 | 709
Completed | 1407 | 697
Not Completed | 17 | 12
Not completed — Lost to Follow-up | 12 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Serious Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV | Total
Number analyzed (Participants) | 1424 | 709 | 2133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1424 | 709 | 2133
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Weeks] | 6.27 (0.280) | 6.30 (0.310) | 6.28 (0.291)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 718 | 356 | 1074
  Male | 706 | 353 | 1059
Region of Enrollment [Number; unit: Participants]
  Philippines | 1424 | 709 | 2133

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroprotection for Anti-Hep Bs, Anti-PRP, Anti-Tetanus, and Anti-Diphtheria Antibodies After Vaccination With Either DTaP-Hep B-PRP~T Concomitantly With OPV or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Seroprotection was assessed by means of radioimmunoassay (RIA) for anti-Hepatitis B (Hep Bs) and anti-PRP antibodies, enzyme immunoassay (EIA) for anti-Tetanus, and serum neutralization (SN) for anti-Diphtheria.
  Seroprotection was defined as titers ≥ 10 mIU/mL for anti-Hep Bs; ≥ 0.15 μg/mL for anti-PRP; ≥ 0.01 IU/mL for anti-Tetanus and anti-Diphtheria at 30 days after the third vaccination.
Time Frame: 1 month post third vaccination
Population: Seroprotection was assessed in a subset of participants available for the endpoint, the per-protocol population.
Measure: Number; unit: Participants
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received 3 doses of the DTaP-Hep B-PRP~T concomitantly with OPV vaccine, 1 dose each at 6, 10, and 14 weeks of age.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received 3 doses of Tritanrix-Hep B/ Hib™ concomitantly with OPV vaccines at 6, 10 and 14 weeks of age.
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 246 | 123
Participants
  Anti-Hep Bs (N = 246, 122) | 239 | 119 [0 to 0]
  Anti-PRP (N = 218, 122) | 210 | 121 [0 to 0]
  Anti-Diphtheria (N = 246, 123) | 217 | 109 [0 to 0]
  Anti-Tetanus (N = 246,123) | 246 | 123 [0 to 0]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Vaccine Antibodies After Vaccination With Either DTaP-Hep B-PRP-T Concomitantly With OPV or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Immunogenicity was assessed by means of radioimmunoassay (RIA) for anti-Hepatitis B (Hep Bs) and anti-PRP antibodies; enzyme immunoassay (EIA) for anti-Tetanus; serum neutralization (SN) for anti-Diphtheria; and enzyme-linked immunosorbent assay (ELISA) for anti-Pertusiss (PT) and anti-Filamentous Hemagglutinin (FHA) titers at Day 150, 1 month after the third vaccination.
Time Frame: 1 month post third vaccination
Population: GMTs were assessed in a subset of the participants available for the endpoint, the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Group 1: DTaP-Hep B-PRP-T + OPV: Participants received 3 doses of the DTaP-Hep B-PRP-T Concomitantly with OPV vaccine, 1 dose each at 6, 10, and 14 weeks of age.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received 3 doses of Tritanrix-Hep B/Hib™ Concomitantly with OPV vaccine, 1 dose each at 6, 10, and 14 weeks of age.
Arm/Group | Group 1: DTaP-Hep B-PRP-T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 246 | 123
Titers
  Anti-Hep Bs (N = 246, 122) | 464 [380 to 567] | 343 [265 to 444]
  Anti-PRP (N = 218, 121) | 3.02 [2.47 to 3.69] | 10.3 [8.30 to 12.8]
  Anti-Diphtheria (N = 246, 123) | 0.025 [0.022 to 0.028] | 0.023 [0.019 to 0.028]
  Anti-Tetanus (N = 246, 123) | 1.05 [0.958 to 1.14] | 1.31 [1.14 to 1.49]
  Anti-Pertusiss (N = 245, 108) | 139 [127 to 152] | 81.5 [57.3 to 116]
  Anti-Filamentous Hemagglutinin (N = 205, 94) | 86.7 [80.0 to 93.9] | 9.17 [7.33 to 11.5]

3. Primary Outcome: Number of Participants With Observed High Fever During the 7-Day After Vaccination With DTaP-Hep B-PRP~T Concomitantly With OPV or Tritanrix-Hep B/ Hib™ Concomitantly With OPV.
Description: Occurence of at least one high fever episode (≥ 39.6ºC rectal temperature equivalent) observed within 7 days after any of the three injections.
Time Frame: Day 0 to Day 7 post-vaccination
Population: Safety was assessed on the safety analysis (intent-to-treat) population. Two participants in Group 1 were given the Group 2 vaccine; 3 participants in Group 2 were given the Group 1 vaccine. The data were analyzed and presented according to the actual treatment received and with the total number (N) available for the endpoint at each time-point.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 1425 | 708
Participants
  Post-any Vaccination (N = 1419, 705) | 5 | 8 [0 to 0]
  Post-vaccination 1 (N = 1419, 705) | 3 | 1 [0 to 0]
  Post-vaccination 2 (N = 1408, 698) | 1 | 3 [0 to 0]
  Post-vaccination 3 (N = 1405, 698) | 1 | 4 [0 to 0]

4. Secondary Outcome: Number of Participants Reporting At Least One Solicited Injection Site Reaction or Systemic Reactions Following Each Vaccination With Either DTaP-Hep B-PRP-T Concomitantly With OPV or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Solicited injection site reactions: Pain, Erythema, and Swelling; Solicited systemic reactions; Fever (temperature), Vomiting, Abnormal Crying, Drowsiness, Loss of Appetite, and irritability.
  Grade 3 reactions are defined as: Pain - cries when injected limb is moved; Erythema and Swelling - ≥ 5cm; Fever - rectal temperature ≥ 39.6ºC; Vomiting - ≥6 episodes per 24 hours; Crying - inconsolable crying for >3 hours; Somnolence - sleeping most of the time or difficulty to wake up; Anorexia - refuses ≥3 feeds; and Irritability - inconsolable.
Time Frame: Day 0 to Day 7 after vaccination
Population: Safety was assessed on the safety analysis (intent-to-treat) population. Two participants in Group 1 were given the Group 2 vaccine; 3 participants in Group 2 were given the Group 1 vaccine. The data were analyzed and presented according to the actual treatment received.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 1425 | 708
Participants
  Injection site Pain post any vaccination | 1092 | 636
  Grade 3 Injection site Pain post any vaccination | 344 | 295
  Injection site Pain Post-vaccination 1 | 958 | 573 [0 to 0]
  Injection site Pain Post-vaccination 2 | 751 | 463 [0 to 0]
  Injection site Pain Post-vaccination 3 | 616 | 407 [0 to 0]
  Injection site Erythema Post any vaccination | 794 | 497 [0 to 0]
  Grade 3 Inject. site Erythema Post any vaccination | 16 | 16 [0 to 0]
  Injection site Erythema Post-vaccination 1 | 543 | 353 [0 to 0]
  Injection site Erythema Post-vaccination 2 | 448 | 320 [0 to 0]
  Injection site Erythema Post-vaccination 3 | 408 | 283 [0 to 0]
  Injection site Swelling Post any vaccination | 719 | 503 [0 to 0]
  Grade 3 Inject. site Swelling Post any vaccination | 15 | 35 [0 to 0]
  Injection site Swelling Post-vaccination 1 | 576 | 423 [0 to 0]
  Injection site Swelling Post-vaccination 2 | 438 | 343 [0 to 0]
  Injection site Swelling Post-vaccination 3 | 365 | 288 [0 to 0]
  Fever Post any vaccination | 523 | 394 [0 to 0]
  Grade 3 Fever Post any vaccination | 5 | 8 [0 to 0]
  Fever Post-vaccination 1 | 282 | 248 [0 to 0]
  Fever Post-vaccination 2 | 222 | 165 [0 to 0]
  Fever Post-vaccination 3 | 187 | 156 [0 to 0]
  Vomiting Post any vaccination | 266 | 172 [0 to 0]
  Grade 3 Vomiting Post any vaccination | 2 | 3 [0 to 0]
  Vomiting Post-vaccination 1 | 193 | 118 [0 to 0]
  Vomiting Post-vaccination 2 | 105 | 83 [0 to 0]
  Vomiting Post-vaccination 3 | 72 | 52 [0 to 0]
  Crying post any vaccination | 567 | 381 [0 to 0]
  Grade 3 Crying post any vaccination | 5 | 0
  Crying post-vaccination 1 | 431 | 301
  Crying post-vaccination 2 | 275 | 193
  Crying post-vaccination 3 | 205 | 152
  Somnolence post any vaccination | 673 | 360
  Grade 3 Somnolence post any vaccination | 43 | 35
  Somnolence post-vaccination 1 | 527 | 282
  Somnolence post-vaccination 2 | 368 | 216
  Somnolence post-vaccination 3 | 255 | 150
  Anorexia post any vaccination | 396 | 250
  Grade 3 Anorexia post any vaccination | 10 | 8
  Anorexia post-vaccination 1 | 235 | 159
  Anorexia post-vaccination 2 | 201 | 118
  Anorexia post-vaccination 3 | 130 | 97
  Irritability post any vaccination | 945 | 539
  Grade 3 Irritability post any vaccination | 33 | 32
  Irritability post-vaccination 1 | 823 | 471
  Irritability post-vaccination 2 | 499 | 331
  Irritability post-vaccination 3 | 369 | 266

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 238 post-vaccination.
Description: Two participants in Group 1 were given the Group 2 vaccine; 3 participants in Group 2 were given the Group 1 vaccine. The safety data were analyzed and presented according to the actual treatment received.
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Serious Adverse Events (participants affected / at risk) | 31/1425 | 12/708
Other Adverse Events (participants affected / at risk) | 1092/1425 | 636/708
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=1425) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=708)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenia purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 2 (2)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 9 (9) | 3 (3)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 13 (13) | 5 (5)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Convlusion (Nervous system disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=1425) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=708)
Solicited injection site Pain (General disorders) | 958 | 573
Solicited injection site Erythema (General disorders) | 543 | 353
Solicited injection site Swelling (General disorders) | 576 | 423
Pyrexia (General disorders) | 282 | 248
Vomiting (Gastrointestinal disorders) | 193 | 118
Crying (Psychiatric disorders) | 431 | 301
Anorexia (Metabolism and nutrition disorders) | 235 | 159
Somnolence (Nervous system disorders) | 527 | 282
Upper respiratory tract infection (Infections and infestations) | 481 | 210
Irritability (Psychiatric disorders) | 823 | 471
Rhinitis (Infections and infestations) | 93 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications